CLINICAL TRIAL: NCT06986967
Title: Retrograde Versus Antegrade Perfusion in Low-Moderate Hypothermia for Aortic Arch Surgery
Acronym: ACP vs RCP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Pro00116844
Record Dates: First submitted 2025-04-29; First posted 2025-05-23 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Brain Function; Hemiarch Cardiac Procedure
Keywords: Antegrade Perfusion; Retrograde Perfusion; Brain Perfusion; Circulatory Arrest

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The neuroimaging personnel will be blinded to the assignment of the subject.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1: Antegrade Perfusion (Active Comparator): In antegrade perfusion, the surgeon accesses one of two arteries that branch off from the aorta (the artery that delivers blood to the rest of the body) to provide blood to the brain.
  Interventions: Procedure: Antegrade Perfusion
- Arm 2: Retrograde Perfusion (Active Comparator): In retrograde perfusion, the surgeon accesses the superior vena cava (large vein bringing blood back to the heart) to supply blood to the brain.
  Interventions: Procedure: Retrograde Perfusion

INTERVENTIONS:
Procedure: Antegrade Perfusion — Procedure in which the surgeon accesses one of two arteries that branch off from the aorta to provide blood to the brain.
  Arms: Arm 1: Antegrade Perfusion
Procedure: Retrograde Perfusion — Procedure in which the surgeon accesses the superior vena cava to supply blood to the brain.
  Arms: Arm 2: Retrograde Perfusion

SUMMARY:
The purpose of this study is to compare brain function after surgical circulatory arrest using either antegrade perfusion or retrograde perfusion.

DETAILED DESCRIPTION:
The purpose of this study is to compare brain function after surgical circulatory arrest (surgeon stops the heart-lung machine to work on the heart) in antegrade perfusion versus retrograde perfusion. There are 2 ways to supply blood to the brain, antegrade and retrograde perfusion. In antegrade perfusion, the surgeon accesses one of two arteries that branch off from the aorta (the artery that delivers blood to the rest of the body) to provide blood to the brain. In retrograde perfusion, the surgeon accesses the superior vena cava (large vein bringing blood back to the heart) to supply blood to the brain.

It is standard practice to cool the patient down during this type of surgery to help protect the brain. Despite measures to safeguard brain health, some patients still experience postoperative cognitive decline such as confusion, delirium and agitation. The investigators are conducting this study to see which method of perfusing the brain is superior and decreases the symptoms of confusion, delirium and agitation.

ELIGIBILITY:
Inclusion Criteria:

1. > 18 years of age
2. Participant's that are scheduled for elective proximal aortic reconstructive surgery (ascending aorta + aortic valve or root) with concomitant proximal hemi-arch replacement via median sternotomy

Exclusion Criteria:

1. < 18 years of age
2. history of symptomatic cerebrovascular disease, e.g., prior stroke with residual deficit
3. current alcoholism (> 2 drinks/day)
4. current psychiatric illness requiring pharmacotherapy
5. current drug abuse (any illicit drug use in the past 3 months)
6. hepatic insufficiency (liver function tests > 1.5 times the upper limit of normal)
7. severe pulmonary insufficiency (requiring home oxygen therapy)
8. renal failure (serum creatinine > 2.0 mg/dL)
9. claustrophobic fear
10. unable to read and thus unable to complete the cognitive testing
11. pregnant women
12. patients who score <19 om the Montreal Cognitive Assessment (MoCA) or ≥27 on the baseline Center for Epidemiological Studies Depression (CES-D) scale
13. patients who have pre-existing unsafe implants for 3 Tesla magnetic resonance imaging (MRI)
14. Patients who have received chemotherapy in the last 12 months or radiation to the brain

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-04-18 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Change in neurocognitive function as measured by the Montreal Cognitive Assessment (MoCA) | Baseline to 4 weeks
  The MoCA is a brief screening tool used to assess cognitive function. It consists of 30 tasks covering various cognitive domains, including attention, memory, visuospatial abilities, and executive function. The total score ranges from 0 to 30, where a higher score indicates better cognitive function.

SECONDARY OUTCOMES:
Effect of Antegrade Perfusion (ACP) vs Retrograde Perfusion (RCP) on brain white matter patency | Baseline, prior to discharge from hospital (up to 7 days), and at 4 weeks
  Measured by MRI at baseline, prior to discharge, and at 4 weeks.
Effect of Antegrade Perfusion (ACP) vs Retrograde Perfusion (RCP) on functional connectivity | Baseline and at 4 weeks
  Measured by MRI at baseline and at 4 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Mathew, M.D., Study Chair — Duke University
Locations (1):
- Duke Univeristy, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes